CLINICAL TRIAL: NCT02655822
Title: A Phase 1/1b, Open-Label, Multicenter, Repeat-Dose, Dose-Selection Study of Ciforadenant as Single Agent and in Combination With Atezolizumab in Patients With Selected Incurable Cancers
Brief Title: Phase 1/1b Study to Evaluate the Safety and Tolerability of Ciforadenant Alone and in Combination With Atezolizumab in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corvus Pharmaceuticals, Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-444-001
Record Dates: First submitted 2016-01-08; First posted 2016-01-14 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-07

CONDITIONS: Renal Cell Cancer; Metastatic Castration Resistant Prostate Cancer
Keywords: RCC; Kidney Cancer; mCRPC; Prostate Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Prostatic Neoplasms | interventions — ciforadenant; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 - Closed (Experimental): Ciforadenant
  Interventions: Drug: Ciforadenant
- Cohort 2 - Closed (Experimental): Ciforadenant
  Interventions: Drug: Ciforadenant
- Cohort 3 - Closed (Experimental): Ciforadenant
  Interventions: Drug: Ciforadenant
- Cohort 4 (Experimental): Ciforadenant + atezolizumab
  Interventions: Drug: Ciforadenant + atezolizumab
- Cohort 5 - Closed (Experimental): Ciforadenant
  Interventions: Drug: Ciforadenant

INTERVENTIONS:
Drug: Ciforadenant — 100 mg orally twice daily for the first 14 days of each 28-day cycle.
  Arms: Cohort 1 - Closed
Drug: Ciforadenant — 100 mg orally twice daily for 28 days of each 28-day cycle.
  Arms: Cohort 2 - Closed
Drug: Ciforadenant — 200 mg orally once daily for the first 14 days of each 28-day cycle.
  Arms: Cohort 3 - Closed
Drug: Ciforadenant + atezolizumab — Ciforadenant 100 mg orally twice daily in combination with atezolizumab intravenously.
  Arms: Cohort 4
Drug: Ciforadenant — Start with 150mg orally twice daily for 28-day cycles; then, increase increments by 100mg/day for 6 dose levels.
  Arms: Cohort 5 - Closed

SUMMARY:
This is a phase 1/1b open-label, multicenter, dose-selection study of ciforadenant, an oral small molecule targeting the adenosine-A2A receptor on T-lymphocytes and other cells of the immune system. This trial will study the safety, tolerability, and anti-tumor activity of ciforadenant as a single agent and in combination with atezolizumab, a PD-L1 inhibitor against various solid tumors. Ciforadenant blocks adenosine from binding to the A2A receptor. Adenosine suppresses the anti-tumor activity of T cells and other immune cells.

DETAILED DESCRIPTION:
This is a phase 1/1b open-label, multicenter, dose-selection study of ciforadenant, an oral small molecule targeting the adenosine-A2A receptor on T-lymphocytes and other cells of the immune system. This trial will study the safety, tolerability, and anti-tumor activity of ciforadenant as a single agent and in combination with atezolizumab, an intravenous PD-L1 inhibitor. Ciforadenant blocks adenosine from binding to the A2A receptor. Adenosine suppresses the anti-tumor activity of T cells and other immune cells.

ELIGIBILITY:
Renal Cell Carcinoma Inclusion Criteria

1. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
2. Documented pathologic diagnosis of clear cell RCC.
3. Relapsed or refractory to 1-2 prior lines of therapy containing at least an anti-PD-(L)1 agent.
4. Measurable disease according to RECIST v1.1
5. Mandatory newly collected tumor biopsy sample obtained prior to treatment initiation.

Renal Cell Carcinoma Exclusion Criteria

1. History of severe hypersensitivity reaction to monoclonal antibodies.
2. Has immunodeficiency or requires treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressant medication during study treatment.
3. Has an active autoimmune disease requiring systemic treatment with in the past 2 years OR a documented history of clinically severe autoimmune disease.

Metastatic Castration-Resistant Prostate Cancer Inclusion Criteria

1. Documentation of disease: progressive CRPC with histologically or cytologically confirmed adenocarcinoma of the prostate.
2. Patients must have radiologically evident metastatic disease, but it can be measurable or non-measurable disease:

   * Measurable disease: nodal, visceral, or extra nodal lesions according to RECIST v1.1 using a diagnostic computed tomography
   * Non-measurable disease: bone only disease (up to 1/3 of study population) per PCWG3 criteria
3. 1-3 prior lines of therapy, including at least one newer generation androgen synthesis inhibitor (e.g., abiraterone) or androgen receptor antagonist (e.g., enzalutamide, apalutamide, darolutamide).
4. Mandatory newly collected tumor biopsy sample obtained prior to treatment initiation.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.

Metastatic Castration-Resistant Prostate Cancer Exclusion Criteria

1. Has pure small-cell histology and variants with predominant (≥ 50%) neuroendocrine differentiation.
2. Has a history of severe hypersensitivity reaction to monoclonal antibodies.
3. Has immunodeficiency or requires treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment or anticipation of need for systemic immunosuppressant medication during study treatment.
4. Has an active autoimmune disease requiring systemic treatment with in the past 2 years OR a documented history of clinically severe autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2016-01; Primary Completion 2021-06 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) of ciforadenant as a single agent and in combination with atezolizumab | 28 days following first administration of ciforadenant
Objective response rate per RECIST v1.1 criteria of ciforadenant as a single agent and in combination with atezolizumab | From start of treatment to end of treatment, up to 72 months
Incidence of treatment-emergent adverse events, as assessed by NCI CTCAE v.4.03, of ciforadenant as a single agent and in combination with atezolizumab | Continuously, up to 72 months
Mean and median Area under the curve (AUC) of ciforadenant | Up to 12 months
Mean and median Maximum concentration (Cmax) of ciforadenant | Up to 12 months
Identify the MDL (maximum dose level) of single agent ciforadenant | From start of treatment to end of treatment, up to 72 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Mobasher, MD, MPH, Study Director — Corvus Pharmaceuticals
Locations (20):
- United States (15):
  - University of Arizona Cancer Center, Tucson, Arizona
  - University of California - San Francisco, San Francisco, California
  - Stanford Cancer Institute, Stanford, California
  - Yale University, New Haven, Connecticut
  - University of Miami Hospital and Clinics, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center Cancer Center, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Monash Health, Clayton, Victoria
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario